CLINICAL TRIAL: NCT01796028
Title: A Multicentric, Randomized, Phase II Study Evaluating the Combination of METFORMIN With TAXOTERE®+Metformine Placebo Versus TAXOTERE®+Metformin for the Treatment of Metastatic Hormone-refractory Prostate Cancer.
Brief Title: Metformin-Docetaxel Association in Metastatic Hormone-refractory Prostate Cancer
Acronym: TAXOMET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-000530-19; 2010/35 (Registry Identifier: TAXOMET)
Record Dates: First submitted 2012-11-12; First posted 2013-02-21 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-01

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A : TAXOTERE® + Metformin placebo (Placebo Comparator): Docetaxel (TAXOTERE®) will be administered at 75 mg/m2. Metformin (or placebo) is formulated into 850 mg tablets for oral administration and is to be dispensed twice a day on a continuous daily dosing schedule
  Interventions: Drug: Placebo; Drug: TAXOTERE®
- Arm B : TAXOTERE® + Metformin (Experimental): Docetaxel (TAXOTERE®) will be administered at 75 mg/m2. Metformin is formulated into 850 mg tablets for oral administration and is to be dispensed twice a day on a continuous daily dosing schedule
  Interventions: Drug: METFORMIN; Drug: TAXOTERE®

INTERVENTIONS:
Drug: METFORMIN
  Other Names: GLUCOPHAGE
  Arms: Arm B : TAXOTERE® + Metformin
Drug: Placebo
  Arms: Arm A : TAXOTERE® + Metformin placebo
Drug: TAXOTERE®

SUMMARY:
Prostate cancer is the second leading cause of mortality in men, representing 10 deaths about of 100 cancers (INVS 2009). Treatment for metastatic prostate cancer, when becoming resistant to hormone-treatment, is mostly resumed to a relatively ineffective chemotherapy (Docetaxel/TAXOTERE®) (1). Recently, numerous clinical and preclinical works showed that Metformin could represent an excellent candidate for treatment of advanced prostate cancer. This is a widely prescribed drug, for type 2 diabetes, with clinical advantage of exhibiting very rare serious side effects. On the other hand, the use of this molecule in patients was associated with a decrease of tumors incidence, in particular prostate cancer (2). Numerous in vitro and in vivo studies support its role as an anti-cancer drug, in several cell lines (3). These experimental results are consistent with a clinical trial pilot study, performed in colorectal cancer, showing anti proliferative effect of Metformin (4). In the field of prostate, F. Bost in J.F. Tanti's team (INSERM U895, Nice) demonstrated that Metformin inhibits cell viability of human prostate cancer cells, via mTOR downregulation and decrease tumor growth in a xenograft model (5). Furthermore, preclinical data performed by this team showed that Metformin increased significantly apoptosis induced by TAXOTERE®. Therefore, by targeting specifically cancer cell metabolism, Metformin offers new promising therapeutic strategy.

The primary objective of this randomized study is to evaluate the biological efficacy of Metformin combination with TAXOTERE® in patients with metastatic hormone-refractory prostate cancer. To achieve this purpose, PSA response rate will be evaluated according to ASTRO definitions (Bubley, Carducci et al. 1999). Concurrently, secondary endpoints will be under investigation in order to evaluate the clinical response according to RECIST criteria, the overall and free-progression survival and the quality of life. Toxicity assessment will also be performed regarding to this drug combination.

Considering the well tolerability of Metformin and the first clinical and pre-clinical data reports of it use in cancer treatment, combining Docetaxel (TAXOTERE®) with Metformin may represent a promising strategy for treatment of hormone-refractory prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer: the current issues In developed countries, prostate cancer represents a major health issue and its incidence is rising globally, due to an aging society (Ferlay, Autier et al. 2007; Damber and Aus 2008). Indeed, over 70% of patients with prostate cancer are over the age of 65 years (Quinn and Babb 2002). In France, prostate cancer is the second most common cause of death from cancer in men and represents 10 deaths about of 100 by cancer (INVS 2009).

Although the screening and early detection have improved, a significant percentage of men diagnosed with prostate cancer will develop metastasis, reducing dramatically the 5-year relative survival (Jemal, Thun et al. 2008).

For patients with metastatic prostate cancer, the first-line treatment relies on androgen suppression following medical therapy or surgical orchiectomy. In about 80 percent of men, androgen ablation leads to symptomatic improvement; however, despite this treatment, the risk of relapse is at a median period of 24 months following hormone manipulation and the survival median is at about 3 years (1995; Sharifi, Dahut et al. 2005).

Clinical management of Castration-Resistant Prostate Cancer:

Currently, treatment for metastatic prostate cancer, when becoming unresponsiveness to androgen deprivation therapy, is mostly resumed to a relatively ineffective chemotherapy. Indeed, this disease state is considered the final stage of the disease in which the morbidity and mortality outlook is extremely bleak, and therapeutic options remain only palliative.

Combined Docetaxel (TAXOTERE®) and prednisone is currently considered the standard of care for men with castration-resistant prostate cancer and detectable metastatic disease, based largely on the simultaneous publication in October 2004 of two larges randomized controlled trials: SWOG 9916 et TAX 327, comparing this combination with the previous established standard of Mitoxantrone and prednisone (Petrylak, Tangen et al. 2004; Tannock, de Wit et al. 2004). While the use of Mitoxantrone led to pain reduction and quality of life improvement, without survival improvement (Tannock, Osoba et al. 1996), Docetaxel became the only approved systemic agent that has been shown to improve overall survival in conjunction with palliative benefits.

Docetaxel (TAXOTERE®) use was based on its ability to induce microtubules polymerization and on the discovery of Bcl-2 expression, an antiapoptotic protein, in prostate cancer cell line from metastatic hormone resistant patients. Indeed, this taxane by phosphorylating Bcl-2 induced apoptosis in cells expressing the protein (McDonnell, Navone et al. 1997).

In the phase III TAX-327 study, median survival was 18.9 month in the 3-week Docetaxel plus prednisone group and 16.5 month compared with mitoxantrone plus prednisone group. Correspondingly, clinically apparent improvements were also reported in terms of PSA response rate, pain response and quality of life, despite the increase in toxicity in the group that received Docetaxel. However, most adverse events associated with Docetaxel were of low grade and were bothersome rather than life-threatening (Tannock, de Wit et al. 2004). In this study, the median duration of the PSA response ranged from 7.7 and 8.2 months and did not differ significantly among the Docetaxel or Mitoxantrone group. In addition, the most common manifestations of metastatic prostate cancer, bone mestastasis that occurs in 65 to 75% (Bubendorf, Schopfer et al. 2000; Roudier, True et al. 2003) are also difficult to quantify accurately. Thus, in prostate cancer, PSA-based endpoint is used to surrogate clinical benefit and demonstrate drug activity in clinical trial.

However, regarding the limited and modest gains of Docetaxel based chemotherapy, trials are now focusing on improving the efficacy of Docetaxel by combining it with novel biological agents, but to date without demonstrable improvements (Ramsay and Leung 2009; Singh, Yam et al. 2010).

Interest of the associate Docetaxel (TAXOTERE®) with Metformin in Hormone-Refractory Prostate Cancer Metformin (N',N'-dimethylbiguanide) is a wildly used anti-diabetic drug which has the clinical advantage of having few side effects except rare lactic acidosis in patients with renal insufficiency (Lalau and Race 1999). Metformin is very effective in treating disorders marked by insulin-resistance. Several recent publications have shown that Metformin has anti-cancer properties

Epidemiologic and clinical evidences:

Several retrospective epidemiologic studies, in diabetic patients, showed that Metformin was associated with reduced risk of all cancer types (Evans, Donnelly et al. 2005; Currie, Poole et al. 2009). Thus, in a first retrospective cohort study of 62,809 type 2 diabetic patients treated in UK, the authors examined the risk of development of solid tumors in relation to treatment with oral agents, human insulin and insulin analogues. Results showed that people on insulin or sulfonylurea were more likely to develop solid cancers than those on Metformin. In this study, Metformin use was associated with lower risk of cancer of the colon or pancreas, but did not seem to affect the risk of breast or prostate cancer (Currie, Poole et al. 2009).

In another UK observational cohort study, cancer was diagnosed among 7.3% of 4,085 Metformin users compared with 11.6% of 4,085 diabetic comparators who had never used Metformin. After adjusting for baseline characteristics, there was still a significantly reduced risk of cancer associated with Metformin (37% lower than the non Metformin users group)(Libby, Donnelly et al. 2009).

In addition to these studies on all cancers, specific investigations reported that Metformin use was also associated with a significant decrease in the relative risk of specific cancers such as pancreatic cancer (Li, Yeung et al. 2009), hepatocellular carcinoma (Donadon, Balbi et al. 2010; Hassan, Curley et al. 2010), prostate (Wright and Stanford 2009) and breast cancers (Bodmer, Meier et al. 2010). Furthermore, in later years of follow up, high doses of Metformin were associated with the greatest reduction in risk of cancer, further supporting a protective effect of Metformin (Evans, Donnelly et al. 2005; Libby, Donnelly et al. 2009) (see review: Beck and Scheen 2010).

Concerning prostate cancer, a Finish and an American study, have shown a significant decrease of prostate cancer incidence in patients treated with Metformin (Murtola, Tammela et al. 2008; Wright and Stanford 2009).

Results from a population-based case-control study in men aged 35-74 years diagnosed with prostate cancer showed that Metformin use was more common in controls than in cases (4,7 versus 2,8%, p = 0,04) (Wright and Stanford 2009), resulting in a 44% risk reduction for prostate cancer.

A recent pilot clinical study, performed on 25 non-diabetic patients, have shown that Metformin reduced significantly the number of colorectal aberrant crypt foci (an endoscopic surrogate marker of colorectal cancer) (Hosono, Endo et al. 2010). This study demonstrates for the first time a beneficial effect of Metformin in anti-cancerous therapy.

Very recent preliminary data, presented at the 33rd Annual San Antonio Breast Cancer Symposium, are consistent with these previous studies showing that Metformin may have beneficial effects on cancer therapy (33rd annual San Antonio Breast Cancer Symposium, December 2010, San Antonio, USA). At the cellular level, combined treatment of metformine and erlotinib led to synergistic growth inhibitory effects in a proliferation assay and a clonogenic assay on breast cancer cells. The combined treatment also robustly reduced activation of EGFR, AKT, ERK and S6 signaling more than when either drug was used alone. Moreover, in a pilot mouse xenograft study, the combination treatment has been shown to shrink tumors by an average of approximately 25% (Meiers PJ 2010). Data from interim safety analysis demonstrated that preoperative metformin, in early stage breast cancer, significantly reduced cancer cell proliferation (as measured by change in Ki67 index) and induced apoptosis (TUNEL, cleaved caspase 3) (Niraula S 2010). Effects of its use was also associated with improved insulin resistance (Niraula S 2010). Those preliminary results showed that meformin was well tolerated with expected mild grade 1 toxicities and no significant QOL effects (Bonanni B 2010; Niraula S 2010). In addition, it has to be noted that no changes in insulin and in glycaemia levels had been reported with metformin use (Bonanni B 2010), except a slight decrease of BMI (Niraula S 2010).

Experimental evidences:

In a xenograft model, Metformin has been shown to inhibit human prostate cancer cell proliferation as well as to decrease significantly tumor growth (Ben Sahra, Laurent et al. 2008). Other investigations demonstrated a direct inhibitory effect of Metformin on the growth of cancer cells originated from breast (Zakikhani, Dowling et al. 2006), ovary (Rattan, Giri et al. 2009), pancreas (Kisfalvi, Eibl et al. 2009) and colon (Buzzai, Jones et al. 2007) as well as on tumor growth in mice models (see review: Ben Sahra, Le Marchand-Brustel et al. 2010)). At the cellular level, Metformin provoked a cell arrest at the G0/G1 stage and induced apoptosis in several cell types.

The mTOR and Akt pathways are frequently activated in cancers, which has been correlated with a poor prognosis. In prostate cancer cells, Tanti's team showed that Metformin strongly inhibited mTOR pathway and down regulated cyclin D1 expression, a protein associated with cellular transformation (Ben Sahra, Laurent et al. 2008). Preclinical preliminary studies, performed in this laboratory, also showed that, combinating Metformin with TAXOTERE®, potentiated significantly the anti-proliferative effect of TAXOTERE®. Furthermore, Metformin also increased TAXOTERE®-induced apoptosis in prostate cancer cells.

2. Location of the work in the context of the current knowledge :

Therefore, by targeting specifically cancer cell metabolism, Metformin offers new promising therapeutic strategies. Indeed, Metformin is very well tolerated and has been used for more than 30 years for the treatment of type II diabetes. The efficiency of Metformin as an anti-proliferative and an anti-tumoral agent in mice and according to recent clinical reports in breast field, raise the possibility that Metformin could be a potential candidate in novel treatment for cancer, especially in human prostate cancer. Here, we hypothesized that Metformin may improve TAXOTERE® efficacy in patient with hormone refractory prostate cancer.

The primary objective of this randomized study is to evaluate the biological efficacy of Metformin combination with TAXOTERE® in patients with metastatic hormone-refractory prostate cancer. To achieve this purpose, PSA response rate will be evaluated according to ASTRO definitions (Bubley, Carducci et al. 1999). Concurrently, secondary endpoints will be under investigation in order to evaluate the clinical response according to RECIST criteria, the overall and free-progression survival and the quality of life. Toxicity assessment will also be performed regarding to this drug combination.

Considering the well tolerability of Metformin and the first clinical and pre-clinical data reports of it use in cancer treatment, combining Docetaxel (TAXOTERE®) with Metformin may represent a promising strategy for treatment of hormone-refractory prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* - Age > 18 years
* Histologically confirmed prostate adenocarcinoma.
* Karnofsky Performance Score > 50%
* Evidence of metastatic disease by the presence of documented locoregional or distant metastases on CT scan of the abdomen and/or pelvis, or bone scintigraphy
* Hormone Resistance Prostate Cancer defined as an increase in PSA level (3 consecutive measurements) after hormonal treatment (surgical castration or androgen blockade)
* No prior chemotherapy (excepted phosphate estramustine or Estracyt®)
* At least one month had to have elapsed between the withdrawal of antiandrogens and enrolment, except LH-RH agonist therapy that must be continued throughout this study.
* Hormonal castration confirmed biologically (testosterone < 0.5 ng/ml)
* Patient with adequate organ function:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Haemoglobin ≥ 9 g/dL
  * Platelets (PTL) ≥ 100 x 109/L
  * AST - ALAT ≤ 2.5x ULN
  * Bilirubin ≤ 1.5 x ULN
  * Creatinine < 150 µmol/l
  * Alkaline phosphatases ≤ 2,5 x ULN
* Patient with life expectancy > 3 months
* Information delivered to patient and informed consent signed by the patient or legal representative
* Patient affiliated with a health insurance system

Exclusion Criteria:

* The patient with at least one of the following criteria could not be included:
* Age < 18 years
* Patient with type II or type I diabetes
* Excessive alcohol intake, acute or chronic.
* Patients already treated with Metformin or an analog
* Known hypersensitivity or allergy to Metformin HCl or any of the excipients.
* Patients with a history of lactic acidosis
* PSA increasement without lesions confirmed by radiography and/or bone scan.
* Testosteronemia > 0.5 ng/ml
* Any radiation within 4 weeks prior to study entry
* Strontium 89 administration within 3 month before inclusion
* Patient with active central nervous system (CNS) metastasis or with history of CNS metastasis
* Peripheral neuropathy with grade > 3 (NCI), unrelated to cancer.
* Patient treated for a cancer other than prostate cancer, with the exception of basal cell carcinoma
* Treatment with any investigational agent
* Treatment on another therapeutic clinical trial within 30 days before enrolment
* Acute or chronic metabolic acidosis
* Patients suffering from severe dehydration
* Permanent contraindication to corticosteroids
* Patient with history of poor compliance or current or past psychiatric conditions or severe acute or chronic medical conditions that would interfere with the ability to comply with the study protocol, such as completion of QoL questionnaire.
* Patient enable to give informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
PSA response rate | Time until main objective analysis is 5 years

SECONDARY OUTCOMES:
Biochemical and clinical progression-free survival | 5 years

OTHER OUTCOMES:
Overall survival: Overall survival will be calculated from the date of randomization to the date of death from any causes. | 5 years
Tolerance of the association: Tolerance will be assessed according to the NCI-CTCAE scale, version 4.0. | 5 YEARS

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc FERRERO, PhD, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre ANTOINE LACASSAGNE, Nice, France

REFERENCES:
- [Derived] Pujalte Martin M, Borchiellini D, Thamphya B, Guillot A, Paoli JB, Besson D, Hilgers W, Priou F, El Kouri C, Hoch B, Deville JL, Schiappa R, Cheli S, Milano G, Tanti JF, Bost F, Ferrero JM. TAXOMET: A French Prospective Multicentric Randomized Phase II Study of Docetaxel Plus Metformin Versus Docetaxel Plus Placebo in Metastatic Castration-Resistant Prostate Cancer. Clin Genitourin Cancer. 2021 Dec;19(6):501-509. doi: 10.1016/j.clgc.2021.08.008. Epub 2021 Sep 17. PMID 34629300
- See also: Related Info — http://www.centreantoinelacassagne.org/